CLINICAL TRIAL: NCT06099925
Title: The Efficacy and Safety of Hetrombopag as Secondary Prevention to Chemotherapy-induced Thrombocytopenia in Patients With Gynecologic Malignancies（the SPRIT TRIAL）
Brief Title: The Efficacy and Safety of Hetrombopag as Secondary Prevention to Chemotherapy-induced Thrombocytopenia in Patients With Gynecologic Malignancies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SYSKY-2023-842-02
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Chemotherapy-induced Thrombocytopenia
MeSH Terms: interventions — hetrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hetrombopag (Experimental): All the 48 patients will be given hetrombopag 5mg/day within 24 hours after chemotherapy
  Interventions: Drug: Hetrombopag

INTERVENTIONS:
Drug: Hetrombopag — All the recruited 48 patients will take hetrombopag 5mg/day within 24 hours after chemotherapy

SUMMARY:
Chemotherapy is an important treatment strategy for gynecological malignancies, such as ovarian cancer, advanced endometrial cancer, cervical cancer. Chemotherapy-induced thrombocytopenia (CIT) is one of the most common chemotherapy-related hematologic toxicities and can increase the risk of bleeding, prolong hospital stays, increase healthcare costs, and, in severe cases, death. It can lead to a reduction in the intensity of chemotherapy doses, delay the next cycle of chemotherapy, or even termination of treatment, thereby affecting the antitumor effect and adversely affecting the long-term survival of these patients. Literature and our data show that when patients develop grade II or worse CIT, the incidence of grade II and above CIT after the next cycle of chemotherapy is 85-92%. Hetrombopag is one of the thrombopoietin receptor agonist (TPO-RA) that has been studied to explore its role in the treatment and prevention of CIT in multiple solid tumors. In order to find out the secondary prevention efficacy of CIT, it is planned to carry out this single-arm prospective study by recruiting 48 patients with gynecological malignancies with grade II CIT or above after chemotherapy, whose platelets has returned to normal after the routine clinical intervention, and then plan to have the next cycle of chemotherapy. The intervention strategy is taking hetrombopag 5mg/day within 24 hours after chemotherapy, then observe the incidence rate of grade II CIT. The endpoint of this study is to assess the effectiveness and safety of hetrombopag for preventing CIT in patients with gynaecological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Pathological diagnosis of gynecological malignancies such as ovarian cancer, cervical cancer, endometrial cancer, etc.
3. Grade 2 or above thrombocytopenia occurred after the previous cycle of chemotherapy, and the platelet count recovered to ≥100×109/L through routine clinical intervention.
4. Patients plan to receive at least one cycle of chemotherapy containing platinum and paclitaxel.
5. Eastern Cooperative Oncology Group Physical Score(ECOG PS) : 0-2.
6. Estimated survival≥ 12 weeks.

Exclusion Criteria:

1. Have received pelvic, spinal radiotherapy and bone field irradiation within 3 months before screening.
2. Grade I and above thrombocytopenia caused by other diseases within 6 months before screening, including but not limited to chronic liver disease, hypersplenism, infection and bleeding,or hematopoietic system diseases .
3. Clinical manifestations of severe bleeding within 2 weeks before screening, including but not limited to gastrointestinal or central nervous system bleeding.
4. Abnormal liver function: patients without liver metastases, Alanine aminotransferase（ALT）/aspartate aminotransferase（AST）>3 upper limit of normal value (ULN); Patients with liver metastases, Alanine aminotransferase（ALT）/aspartate aminotransferase（AST) ≥5 upper limit of normal value (ULN).
5. Abnormal renal function: serum creatinine ≥ 1.5upper limit of normal value (ULN).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-10-16 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
efficacy of hetrombopag | from the date of recruitment to the time of 14 days
  incidence of thrombocytopenia according to Common Terminology Criteria for Adverse Events 5.0(CTCAE5.0)

SECONDARY OUTCOMES:
reduction of dose | from the date of recruitment to the time of 3 weeks
  the percentage of dose reduction due to thrombocytopenia
adverse reactions | from the date of recruitment to the time of 3 weeks
  Incidence of adverse reactions